CLINICAL TRIAL: NCT04571073
Title: Manual Therapy Informed by the Fascia Distortion Model for Plantar Heel Pain: Results of a Single-arm Prospective Effectiveness Study
Brief Title: Recovery From Plantar Heel Pain Using the Fascial Distortion Model a Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisenhower Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joshua D Boucher, Primary Investigator, Eisenhower Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDEAMC17005
Record Dates: First submitted 2020-09-23; First posted 2020-09-30 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Plantar Fasciitis of Both Feet

STUDY DESIGN:
Masking Description: The AI taking the ultrasound images was blinded to study phase of the participant he was screening.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): The only arm in the study was the intervention arm as this is a pilot study.
  Interventions: Procedure: Fascial Distortion Model

INTERVENTIONS:
Procedure: Fascial Distortion Model — Using physical exam and manual manipulation skills informed by the FDM, he identified and treated locations of presumed fascial distortion about the plantar area of the foot; "distortions" could include any of the six reported fascial anomalies in the FDM: continuum distortions, trigger bands, herniated trigger points, folding distortions, cylinder distortions, and tectonic fixations. Each distortion is associated with a recommended reparative manipulation. The purported mechanism of action is that the distortion-specific manipulation restores normal fascial homogeneity.
  Other Names: FDM

SUMMARY:
To assess feasibility and determine preliminary efficacy of Fascial Distortion Model (FDM) for plantar heel pain (PHP) in a pilot study. The FDM is a hands on direct technique that is non-invasive and has been shown in preliminary studies to be effective in treating musculoskeletal (MSK) injuries. Study participants will be Active Duty Service Members (SM) in the Fort Gordon catchment area.

DETAILED DESCRIPTION:
This prospective, single arm pilot study was approved by the Dwight D. Eisenhower Army Medical Center human subjects Institutional Review Board. Participants were recruited from Dwight D. Eisenhower Army Medical Center from March 2018 to February 2019.

Visit 1-Screening and treatment visit The research staff will review the informed consent with potential research participant(s) and will answer any questions the participant may have about the information in the informed consent. Participants that are willing to participate and sign the informed consent will be eligible to be screened for the study. Participants will be provided copies of their signed informed consent.

Participants will be screened for eligibility to participate in the study based on the inclusion/exclusion criteria and their understanding and acceptance of possible side effects that will be clearly identified in the consent form. Participants must have a current history of PHP and be an Active Duty SM. Participants will be required to have provide detailed information on the quantity of pain medications they consume daily and have a stable history of PHP for at least 30 days prior to the start of screening and treatment.

The inclusion and exclusion criteria will be reviewed with the participant to assure the participant meets the criteria required for participation in the study. Initially, participants who meet the study criteria will screened and treatment on day one. During screening, participants will provide or update a demographics questionnaire, Foot Health Status Questionnaire (FHSQ), medication history, medical history information including history of PHP and events leading up to the diagnosis, profile history, and will undergo a musculoskeletal exam and a general physical exam, including vital signs. The involved foot/feet will be undergo ultrasonography to and a thickness of the fascia will be measured via ultrasound. Medication history includes any and all medications currently taking including vitamins and minerals.

Prior to treatment the patient will be seated for at least 30-60 minutes and provide a visual analogue scale (VAS) measurement of their pain at rest, first step, one and two foot jump, squat, walk, and run.

The participant will meet with a provider educated in the FDM who will follow the protocols for treatment of the plantar heel pain to include diagnosis and treatment of: Continuum distortions, trigger bands, herniated trigger points, folding distortions, cylinder distortions, and tectonic fixations. These treatment may/can start in the foot and extend up the lower leg and may involve treatment of decreased range of motion in the foot, ankle, or lower extremity.

The participant will be instructed to not apply heat to the area for the next 48 hours, maintain profile (if they have one) status, and continue to limit their activity as to not re-injure the foot/feet. The participant will return in two to seven days following the treatment.

Visit 2-Second intervention At Visit 2 which will occur at two to seven days, the inclusion and exclusion criteria will be reviewed with the participant to assure the participant continues to meet the criteria required for participation in the study. Patient will report on their activities since the last treatment and if they applied heat to the affected area.

Participants will provide or update a demographics questionnaire, FHSQ, medication history, medical history, profile history, any adverse reactions to prior treatment, and will undergo a musculoskeletal exam and a general physical exam, including vital signs with body mass index.

Prior to treatment the patient will be seated for at least 30-60 minutes and provide a VAS measurement of their pain at rest, first step, one and two foot jump, squat, walk, and run.

The participant will meet with the same provider as during visit one. The provider educated with the FDM will follow the protocols for treatment of the plantar heel pain to include diagnosis and treatment of continuum distortions, trigger bands, herniated trigger points, folding distortions, cylinder distortions, and tectonic fixations. These treatment may/can start in the foot and extend up the lower leg and may involve treatment of decreased range of motion in the foot, ankle, or lower extremity.

The participant will return for last visit at 4 months.

Visit 3 Follow-up, final visit Upon returning for the 4 month follow up, the participant will undergo an exit neurological exam, physical exam, concomitant medications will be reviewed and updated. Participants will provide a FHSQ, and updates to their profile, and any adverse reactions to prior treatment. Ultrasound will be performed to measure the thickness of the plantar fascia by the same provider that measure the fascia on the first visit. Participant will be seated for at least 30-60 minutes and provide a VAS measurement of their pain at rest, first step, one and two foot jump, squat, walk, and run.

Study Termination

The research team may terminate this study at any time and for any reason. If a participant is withdrawn or the study is terminated, investigators will initiate participant intervention according to institutional standard of care procedures. Participants will be terminated from the study for any one of the following reasons:

Withdrawal of informed consent Failure to continue to meet inclusion criteria, meet any of the exclusion criteria or withdrawal by investigator Lost to follow up Serious Adverse event Protocol non compliance Completion of the study

Procedures for early termination:

Update medical history & medication history, Perform physical and musculoskeletal exams, if possible Document reported and/or observed adverse events VAS, FHSQ questionnaire, profile duration, ultrasound plantar fascia thickness measurement completed, if possible

Intervention with the fascial distortion model will be the research procedure, it will be performed by the primary investigator (PI) or a trained member of the research team with direct supervision of the PI.

Instructions for performing the FDM:

Diagnose the correct distortion, one of six options: herniated trigger point (HTP), continuum distortion (CD), trigger band (TB), cylinder distortion (Cyd), folding distortion (FD), and tectonic fixation (TF).

Diagnosis made by patients body language HTP: participant pushes two fingers into the tissues CD: participant pushes with one finger into the tissue on a bony prominence TB: participant sweeping fingers along the tissues in a linear pathway CyD: broad sweeping of tissues or repetitive squeezing FD: holding or cupping the tissues TF: moving tissues/joint through range of motion

Treatment will depend on the diagnosis made HTP: Apply direct firm pressure with the distal phalanx of the first digit into the most tender portion of the tissues in the HTP for five to ten seconds CD: Apply direct firm pressure with the distal phalanx of the first digit through the tissues readjusting to find the most tender position and hold the position for five to thirty seconds.

TB: Apply direct firm pressure with the distal phalanx along the linear plane of tissue drawn out by the patient CyD: Apply direct firm pressure with the distal phalanx of both hands spreading the tissues apart, or apply a cupping device to the tissues, or grab the tissues with the hands and twist the tissues in opposing directions as the PI deems appropriate.

FD: Find the direction in which the fascia is torqued by pulling or pushing in different planes and then once that direction is found, apply traction in that plane that is constant and then quickly add a thrust in the same direction. TF: Find the direction in which the fascia is fixated and move the tissues through the range of motion while applying traction.

Only HTP, CD, and TBs are expected to be discovered and treated throughout the study.

Data Collection:

Participants will be screened on-site at DDEAMC for general inclusion/exclusion criteria. They will be given a full description of the study procedures and asked to read and sign an IRB-approved informed consent form.

Screening and treatment of DDEAMC recruited participants will occur on the DDEAMC outpatient clinic after the participants have been given a full description of the study procedures and have signed a IRB approved consent.

The screening will include: Background information including medical+plantar heel pain+medication histories, inclusion & exclusion criteria evaluation, MSK and physical exams, vital signs, as well as a series of questionnaires listed below.

Study Documentation Data for this trial will be primarily collected in an electronic data capture (EDC). This will be done with DoD AHTLA. It is the investigator's responsibility for the collection and reporting of all clinical and safety data entered and confirm the data is accurate, authentic, attributable, complete, and consistent. The investigator or sub investigator must sign the note in AHLTA to attest the information contained is true and causality of any safety information has been assessed.

The following information will be collected throughout the study at all three encounters:

Physical Exam Vital Signs Medical History PHP History Medication History Update Medications Collect Adverse Events FHSQ VAS Profile status Ultrasound measured plantar fascia thickness at visit one and three

MSK and physical Examinations. A delegated physician AIs will examine the patient for any detectable abnormalities of the following body systems: general appearance; neck; head, eyes, ears, nose, and throat; lungs; heart/cardiovascular; abdomen; neurologic; extremities; back; musculoskeletal; lymphatic; skin; and other. The MSK examination will assess active and passive range of motion, reflexes, sensory, muscle strength with focus on the lower extremities. After the participant had been at rest for 30 minutes pain will be assessed at rest, first step, one and two foot jump, squat, walk, and run.

Vital Signs. Vital signs with body mass index will be measured at screening, Visit 1, and each subsequent office visit. Systolic and diastolic blood pressure and pulse rate over 30 seconds should be taken after patients have been at rest (seated) for at least 2 minutes. Blood pressure should be recorded in mmHg. Pulse rate should be measured in beats per minutes. Weight will be recorded at each office visit and measured in pounds. Height will be taken at screening and measured in inches.

Foot Health Status Questionnaire: The FHSQ is a 29 question questionnaire that is a validated survey with a goodness-of-fit index of 0.9 suggesting a moderate fit of measurement of foot health related to quality of life.

Visual analogue scale (VAS). The VAS will be used to assess the pain at the plantar heel location during rest, first step, one and two foot jump, squat, walk, and run. The participant will plot the pain level along a linear scale that gives a the opportunity for any potential score from zero to one hundred.

Plantar thickness as measured by ultrasound. A trained AI will measure each participant at the beginning of visit one and during visit three with the ultrasound. Measurement will take place just distal to the calcaneus, an image will be saved for each participant and placed in the EDC.

Available subject's data will be used if they withdraw from the project or the research team withdraws them from the project.

Based on other studies related to Fascial Distortion Model and the amount of variables the goal will be to treat 50 feet.

Analysis A per protocol analytic approach using SPSS 26.0 statistical package will be employed to investigate whether manipulation using the FDM for PHP improved outcomes. Descriptive statistics to be performed to describe outcomes at each time point; average value ± standard deviation (SD) will be reported at baseline unless otherwise specified.

Repeated Measures Analysis of Variance (ANOVA) will test the hypothesis that there was a within subject omnibus improvement over time in FHSQ and VAS scores. Statistical assumptions including sphericity to be met. Post-hoc within-subject paired sample t-tests will be used to identify at which time points a statistically significant difference in FHSQ and VAS scores occurred (i.e., at 1- or 16-weeks later relative to baseline). Average values ± standard deviation (SD) will be reported for this analysis. The unit of analysis for both is the participant.

The unit of analysis for plantar fascia thickness is the individual foot, regardless whether one or both feet were treated. A paired sample t-test will compare differences in the thickness of study plantar fascia at 16 weeks post intervention relative to baseline. Given that this is a pilot study, a conventional p-value of ≤ .05 was selected to denote statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military service members
* Ages of 18 to 65 with self-reported heal pain for 30 or more days
* Clinical diagnosis of Plantar heel pain

Exclusion Criteria:

* history of aneurysm
* bleeding disorders
* active cancer
* phlebitis
* thromboembolism
* foot site contraindications (infection, open wound, hematoma, or edema)
* planned deployment within the four months post-screening
* medical condition that would preclude study participation
* pain that would interfere with foot pain reporting.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Foot pain subscale of the Foot Health Status Questionnaire | Change from baseline to 1 week to 4 months
  A validated disease-specific quality of life questionnaire with 19 100-point questions and eight subscales each ranging from 0-100 with higher scores denoting more favorable health status.

SECONDARY OUTCOMES:
Visual analog pain scale (100 point) | Change from baseline to 1 week to 4 months
  Participant marked on a scale from zero (no pain) to severe (extremely painful) for each foot.
Plantar fascia thickness measured by ultrasound | change from baseline to 4 months
  An MSK trained sonographer with MSK radiologist oversight used the same ultrasound machine to obtain the image of the plantar fascia per the approved radiology protocol.
7 other subscales of the Foot Health Status Questionnaire | Change from baseline to 1 week to 4 months
  A validated disease-specific quality of life questionnaire with 19 100-point questions and eight subscales each ranging from 0-100 with higher scores denoting more favorable health status.

OTHER OUTCOMES:
Use of Non steroidal anti-inflammatory medications (NSAID) | change from baseline to 4 months
  A baseline NSAID use was assessed then at future visits it was asked, no change, decreased, or stopped.
Physical profile | change from baseline to 4 months
  A documented Department of the Army Form 3349, or "Physical Profile," the framework used by medical and behavioral health providers to indicate a soldier's functional limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- Dwight D. Eisenhower Army Medical Center, Fort Gordon, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
If I am contacted by another study at that time I will decide whether or not to share the data.

REFERENCES:
- [Background] McMillan AM, Landorf KB, Barrett JT, Menz HB, Bird AR. Diagnostic imaging for chronic plantar heel pain: a systematic review and meta-analysis. J Foot Ankle Res. 2009 Nov 13;2:32. doi: 10.1186/1757-1146-2-32. PMID 19912628
- [Background] Riddle DL, Schappert SM. Volume of ambulatory care visits and patterns of care for patients diagnosed with plantar fasciitis: a national study of medical doctors. Foot Ankle Int. 2004 May;25(5):303-10. doi: 10.1177/107110070402500505. PMID 15134610
- [Background] Uden H, Boesch E, Kumar S. Plantar fasciitis - to jab or to support? A systematic review of the current best evidence. J Multidiscip Healthc. 2011;4:155-64. doi: 10.2147/JMDH.S20053. Epub 2011 May 24. PMID 21655342
- [Background] League AC. Current concepts review: plantar fasciitis. Foot Ankle Int. 2008 Mar;29(3):358-66. doi: 10.3113/FAI.2008.0358. No abstract available. PMID 18348838
- [Background] Lemont H, Ammirati KM, Usen N. Plantar fasciitis: a degenerative process (fasciosis) without inflammation. J Am Podiatr Med Assoc. 2003 May-Jun;93(3):234-7. doi: 10.7547/87507315-93-3-234. PMID 12756315
- [Background] Trojian T, Tucker AK. Plantar Fasciitis. Am Fam Physician. 2019 Jun 15;99(12):744-750. PMID 31194492
- [Background] Buchbinder R. Clinical practice. Plantar fasciitis. N Engl J Med. 2004 May 20;350(21):2159-66. doi: 10.1056/NEJMcp032745. No abstract available. PMID 15152061
- [Background] Zugel M, Maganaris CN, Wilke J, Jurkat-Rott K, Klingler W, Wearing SC, Findley T, Barbe MF, Steinacker JM, Vleeming A, Bloch W, Schleip R, Hodges PW. Fascial tissue research in sports medicine: from molecules to tissue adaptation, injury and diagnostics: consensus statement. Br J Sports Med. 2018 Dec;52(23):1497. doi: 10.1136/bjsports-2018-099308. Epub 2018 Aug 2. PMID 30072398
- [Background] Typaldos S. FDM Clinical and Theoretical Application of the Fascial Distortion Model Within the Practice of Medicine and Surgery. 4th Edition. Typaldos Publishing Co; 2002.
- [Background] Typaldos S. Introducing the Fascial Distortion Model. Am Acad of Osteopath J. 1994. 14-36.
- [Background] Richter D, Karst M, Buhck H, Fink MG. Efficacy of Fascial Distortion Model Treatment for Acute, Nonspecific Low-Back Pain in Primary Care: A Prospective Controlled Trial. Altern Ther Health Med. 2017 Sep;23(5):AT5522. Epub 2017 Jun 23. PMID 28646809
- [Background] Fink M, Schiller J, Buhck H. [Efficacy of a manual treatment method according to the fascial distortion model in the management of contracted ("frozen") shoulder]. Z Orthop Unfall. 2012 Sep;150(4):420-7. doi: 10.1055/s-0032-1314996. Epub 2012 Aug 23. German. PMID 22918828
- [Background] Boucher JD, Figueroa J. Restoration of Full Shoulder Range of Motion After Application of the Fascial Distortion Model. J Am Osteopath Assoc. 2018 May 1;118(5):341-344. doi: 10.7556/jaoa.2018.044. PMID 29507951
- [Background] Schulze C, Finze S, Bader R, Lison A. Treatment of medial tibial stress syndrome according to the fascial distortion model: a prospective case control study. ScientificWorldJournal. 2014;2014:790626. doi: 10.1155/2014/790626. Epub 2014 Oct 14. PMID 25379543
- [Background] Baird CJ, Shumate SM, et al. The Effects of the Fascial Distortion Model on Chronic Hamstring Tightness. Topics in Integrative Health Care. 2014;5(3).
- [Background] Ribar J, Capistrant T. Cranial and Fascial Distortion Techniques Used as Complementary Treatments Alleviate Migraine Headache: A Case Report. American Academy of Osteopathy. 2015; 25(3).
- [Background] James SJ, Hudnall J. Use of the Fascial Distortion Model to Evaluate a Limp in a Child. J Am Osteopath Assoc. 2017 Jun 1;117(6):399-402. doi: 10.7556/jaoa.2017.079. PMID 28556863
- [Background] Palomo-Lopez P, Lopez-Lopez D, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Rodriguez-Sanz D, Fernandez-Carnero J, Martiniano J, Calvo-Lobo C. Concurrent Validity of the Foot Health Status Questionnaire and Study Short Form 36 for Measuring the Health-Related Quality of Life in Patients with Foot Problems. Medicina (Kaunas). 2019 Nov 19;55(11):750. doi: 10.3390/medicina55110750. PMID 31752435
- [Background] Riskowski JL, Hagedorn TJ, Hannan MT. Measures of foot function, foot health, and foot pain: American Academy of Orthopedic Surgeons Lower Limb Outcomes Assessment: Foot and Ankle Module (AAOS-FAM), Bristol Foot Score (BFS), Revised Foot Function Index (FFI-R), Foot Health Status Questionnaire (FHSQ), Manchester Foot Pain and Disability Index (MFPDI), Podiatric Health Questionnaire (PHQ), and Rowan Foot Pain Assessment (ROFPAQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S229-39. doi: 10.1002/acr.20554. No abstract available. PMID 22588747
- [Background] Landorf KB, Twyford GN, Cotchett MP, Whittaker GA. Revised minimal important difference values for the visual analogue scale and Foot Health Status Questionnaire when used for plantar heel pain. J Foot Ankle Res. 2024 Dec;17(4):e70021. doi: 10.1002/jfa2.70021. PMID 39682003
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Mohseni-Bandpei MA, Nakhaee M, Mousavi ME, Shakourirad A, Safari MR, Vahab Kashani R. Application of ultrasound in the assessment of plantar fascia in patients with plantar fasciitis: a systematic review. Ultrasound Med Biol. 2014 Aug;40(8):1737-54. doi: 10.1016/j.ultrasmedbio.2014.03.001. Epub 2014 May 3. PMID 24798393
- [Background] Ahn JH, Lee CW, Park C, Kim YC. Ultrasonographic examination of plantar fasciitis: a comparison of patient positions during examination. J Foot Ankle Res. 2016 Sep 15;9:38. doi: 10.1186/s13047-016-0171-4. eCollection 2016. PMID 27651833
- [Background] Tylpaldos S, Nagel M, et al. The Fascial Distortion Model as Developed by Stephen Tylpaldos. 1st ed. Edina, MN: Beaver Pond Press; c2015
- [Background] About Adult BMI. Center for Disease Control and Prevention website. Updated June 30, 2020. Accessed July 11, 2020. https://www.cdc.gov/healthyweight/assessing/bmi/adult_bmi/index.html
- [Background] Blyth FM, March LM, Nicholas MK, Cousins MJ. Self-management of chronic pain: a population-based study. Pain. 2005 Feb;113(3):285-292. doi: 10.1016/j.pain.2004.12.004. PMID 15661435
- [Background] Chenot JF, Greitemann B, Kladny B, Petzke F, Pfingsten M, Schorr SG. Non-Specific Low Back Pain. Dtsch Arztebl Int. 2017 Dec 25;114(51-52):883-890. doi: 10.3238/arztebl.2017.0883. PMID 29321099
- [Background] Monto RR. Platelet-rich plasma efficacy versus corticosteroid injection treatment for chronic severe plantar fasciitis. Foot Ankle Int. 2014 Apr;35(4):313-8. doi: 10.1177/1071100713519778. Epub 2014 Jan 13. PMID 24419823
- [Background] Landsman AS, Catanese DJ, Wiener SN, Richie DH Jr, Hanft JR. A prospective, randomized, double-blinded study with crossover to determine the efficacy of radio-frequency nerve ablation for the treatment of heel pain. J Am Podiatr Med Assoc. 2013 Jan-Feb;103(1):8-15. doi: 10.7547/1030008. PMID 23328847
- [Background] Shetty SH, Dhond A, Arora M, Deore S. Platelet-Rich Plasma Has Better Long-Term Results Than Corticosteroids or Placebo for Chronic Plantar Fasciitis: Randomized Control Trial. J Foot Ankle Surg. 2019 Jan;58(1):42-46. doi: 10.1053/j.jfas.2018.07.006. Epub 2018 Nov 15. PMID 30448183
- [Background] Franchini M, Cruciani M, Mengoli C, Marano G, Pupella S, Veropalumbo E, Masiello F, Pati I, Vaglio S, Liumbruno GM. Efficacy of platelet-rich plasma as conservative treatment in orthopaedics: a systematic review and meta-analysis. Blood Transfus. 2018 Nov;16(6):502-513. doi: 10.2450/2018.0111-18. Epub 2018 Sep 3. PMID 30201082
- [Background] Chew KT, Leong D, Lin CY, Lim KK, Tan B. Comparison of autologous conditioned plasma injection, extracorporeal shockwave therapy, and conventional treatment for plantar fasciitis: a randomized trial. PM R. 2013 Dec;5(12):1035-43. doi: 10.1016/j.pmrj.2013.08.590. Epub 2013 Aug 22. PMID 23973504
- [Background] Eslamian F, Shakouri SK, Jahanjoo F, Hajialiloo M, Notghi F. Extra Corporeal Shock Wave Therapy Versus Local Corticosteroid Injection in the Treatment of Chronic Plantar Fasciitis, a Single Blinded Randomized Clinical Trial. Pain Med. 2016 Sep;17(9):1722-31. doi: 10.1093/pm/pnw113. Epub 2016 Jun 8. PMID 27282594
- [Background] Thalhamer C. A fundamental critique of the fascial distortion model and its application in clinical practice. J Bodyw Mov Ther. 2018 Jan;22(1):112-117. doi: 10.1016/j.jbmt.2017.07.009. Epub 2017 Jul 25. PMID 29332733
- [Background] Kwong EH, Findley TW. Fascia--Current knowledge and future directions in physiatry: narrative review. J Rehabil Res Dev. 2014;51(6):875-84. doi: 10.1682/JRRD.2013.10.0220. PMID 25356911
- [Background] Bordoni B, Zanier E. Clinical and symptomatological reflections: the fascial system. J Multidiscip Healthc. 2014 Sep 18;7:401-11. doi: 10.2147/JMDH.S68308. eCollection 2014. PMID 25258540
- [Background] Zein-Hammoud M, Standley PR. Modeled Osteopathic Manipulative Treatments: A Review of Their in Vitro Effects on Fibroblast Tissue Preparations. J Am Osteopath Assoc. 2015 Aug;115(8):490-502. doi: 10.7556/jaoa.2015.103. PMID 26214822
- [Background] Swanson RL 2nd. Biotensegrity: a unifying theory of biological architecture with applications to osteopathic practice, education, and research--a review and analysis. J Am Osteopath Assoc. 2013 Jan;113(1):34-52. doi: 10.7556/jaoa.2013.113.1.34. PMID 23329804
- [Background] Rodrigues RN, Lopes AA, Torres JM, Mundim MF, Silva LL, Silva BR. Compressive neuropathy of the first branch of the lateral plantar nerve: a study by magnetic resonance imaging. Radiol Bras. 2015 Nov-Dec;48(6):368-72. doi: 10.1590/0100-3984.2013.0028. PMID 26811554
- [Background] Trescot AM. Peripheral Nerve Entrapments: Clinical Diagnosis and Management. Springer International Publishing; 2016